CLINICAL TRIAL: NCT02108262
Title: A Phase 2b, Multi-center, Randomized, Placebo-controlled, Dose-ranging Study to Investigate the Safety and Tolerability of Multiple Dose Administration of CSL112 in Subjects With Acute Myocardial Infarction.
Brief Title: A Phase 2b Study of CSL112 in Subjects With Acute Myocardial Infarction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-HDL-12-77; 2013-003458-26 (EudraCT Number)
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — CSL112

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CSL112 - low dose (Experimental): CSL112 (low dose) is to be administered as an intravenous (IV) infusion once weekly for 4 consecutive weeks.
  Interventions: Biological: CSL112
- CSL112 - high dose (Experimental): CSL112 (high dose) is to be administered as an IV infusion once weekly for 4 consecutive weeks.
  Interventions: Biological: CSL112
- Placebo (Placebo Comparator): Placebo is to be administered as an IV infusion at the same frequency, volume and duration as either the low dose or high dose CSL112 infusion.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CSL112 — CSL112 is a novel formulation of apolipoprotein A-I (apoA-I) purified from human plasma and reconstituted to form high-density lipoprotein (HDL) particles.
  Arms: CSL112 - high dose; CSL112 - low dose
Biological: Placebo — 0.9% weight/volume sodium chloride solution (ie, normal saline)
  Arms: Placebo

SUMMARY:
This is a multicenter randomized, double-blind, placebo-controlled, parallel-group, dose-ranging phase 2b study to investigate the hepatic and renal safety and tolerability of multiple dose administration of two dose levels of CSL112 compared with placebo in subjects with acute myocardial infarction (AMI).

ELIGIBILITY:
Inclusion Criteria:

* Men or women, at least 18 years of age, with evidence of myocardial necrosis in a clinical setting consistent with a type I (spontaneous) acute myocardial infarction (AMI), in the last week.

Exclusion Criteria:

* Ongoing hemodynamic instability
* Evidence of hepatobiliary disease
* Evidence of chronic kidney disease (CKD) (Stage III, IV, or V), defined as moderate or severe renal impairment or if subject is receiving dialysis
* Evidence of unstable renal function
* History of acute kidney injury after previous exposure to an intravenous contrast agent.
* Known history of allergies, hypersensitivity or deficiencies to CSL112 or any of its components
* Other severe comorbid condition, concurrent medication, or other issue that renders the subject unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1267 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Denise D'Andrea, Study Director — CSL Behring
Locations (189):
- United States (48):
  - Study Site 16101, Birmingham, Alabama
  - Study Site 16078, Huntsville, Alabama
  - Study Site - 16168, Concord, California
  - Study Site 16168, Concord, California
  - Study Site 16147, Sacramento, California
  - Study Site 16022, Torrance, California
  - Study Site 16130, Littleton, Colorado
  - Study Site 16170, Bridgeport, Connecticut
  - Study Site 16135, Danbury, Connecticut
  - Study Site 16148, Clearwater, Florida
  - Study Site 16003, Jacksonville, Florida
  - Study Site 16144, Atlanta, Georgia
  - Study Site 16112, Boise, Idaho
  - Study Site 16060, Evanston, Illinois
  - Study Site 16179, Elkhart, Indiana
  - Study Site 16102, Indianapolis, Indiana
  - Study Site 16025, West Des Moines, Iowa
  - Study Site 16088, Lexington, Kentucky
  - Study Site 16004, Lexington, Kentucky
  - Study Site 16016, Louisville, Kentucky
  - Study Site 16208, Alexandria, Louisiana
  - Study Site 16062, Auburn, Maine
  - Study Site 16079, Bangor, Maine
  - Study Site 16031, Baltimore, Maryland
  - Study Site 16028, Detroit, Michigan
  - Study Site 16061, Petoskey, Michigan
  - Study Site 16211, Minneapolis, Minnesota
  - Study Site 16234, Saint Paul, Minnesota
  - Study Site 16063, Tupelo, Mississippi
  - Study Site 16033, Brooklyn, New York
  - Study Site 16174, Buffalo, New York
  - Study Site 16213, New York, New York
  - Study Site 16056, Durham, North Carolina
  - Study Site 16201, Elizabeth City, North Carolina
  - Study Site 16014, High Point, North Carolina
  - Study Site 16024, Winston-Salem, North Carolina
  - Study Site 16047, Cincinnati, Ohio
  - Study Site 16026, Hershey, Pennsylvania
  - Study Site 16100, Lancaster, Pennsylvania
  - Study Site 16017, Philadelphia, Pennsylvania
  - Study Site 16039, Greenwood, South Carolina
  - Study Site 16018, Rapid City, South Dakota
  - Study Site 16202, Greeneville, Tennessee
  - Study Site 16015, Amarillo, Texas
  - Study Site 16099, Dallas, Texas
  - Study Site 16241, Wichita Falls, Texas
  - Study Site 16038, Richmond, Virginia
  - Study Site 16166, Wausau, Wisconsin
- Australia (5):
  - Study Site 10002, Herston, Queensland
  - Study Site 10005, Adelaide, South Australia
  - Study Site 10012, Woodville South, South Australia
  - Study Site 10006, Epping, Victoria
  - Study Site 10007, Geelong, Victoria
- Austria (3):
  - Study Site 11004, Innsbruck
  - Study Site 11002, Vienna
  - Study Site 11001, Vienna
- Bulgaria (19):
  - Study Site 12005, Blagoevgrad
  - Study Site 12008, Burgas
  - Study Site 12006, Dobrich
  - Study Site 12021, Haskovo
  - Study Site 12009, Pazardzhik
  - Study Site 12019, Pazardzhik
  - Study Site 12016, Pleven
  - Study Site 12014, Plovdiv
  - Study Site 12018, Plovdiv
  - Study Site 12017, Sandanski
  - Study Site 12003, Sofia
  - Study Site 12001, Sofia
  - Study Site 12004, Sofia
  - Study Site 12012, Sofia
  - Study Site 12010, Sofia
  - Study Site 12013, Sofia
  - Study Site 12011, Varna
  - Study Site 12002, Veliko Tarnovo
  - Study Site 12007, Yambol
- Canada (9):
  - Study Site - 13003, Edmonton, Alberta
  - Study Site - 13002, Edmonton, Alberta
  - Study Site - 13017, Penticton, British Columbia
  - Study Site - 13012, Victoria, British Columbia
  - Study Site - 13019, St. John's, Newfoundland and Labrador
  - Study Site - 13008, London, Ontario
  - Study Site - 13010, Newmarket, Ontario
  - Study Site - 13014, Montreal, Quebec
  - Study Site - 13007, Québec
- Czechia (16):
  - Study Site 14010, Brno
  - Study Site 14006, Brno
  - Study Site 14004, Hradec Králové
  - Study Site 14012, Jablonec nad Nisou
  - Study Site 14011, Jihlava
  - Study Site 14016, Kolín
  - Study Site 14017, Náchod
  - Study Site 14007, Ostrava
  - Study Site 14003, Pardubice
  - Study Site 14002, Prague
  - Study Site 14001, Prague
  - Study Site 14015, Prague
  - Study Site 14009, Prague
  - Study Site 14008, Praha 4 - Krc
  - Study Site 14014, Teplice
  - Study Site 14005, Ústí nad Orlicí
- Denmark (5):
  - Study Site 15001, Aalborg
  - Study Site 15005, Esbjerg
  - Study Site 15002, Hellerup
  - Study Site 15004, Hvidovre
  - Study Site 15003, Odense
- France (6):
  - Study Site - 25003, Pessac, Gironde
  - Study Site - 25005, Toulouse, Haute Garonne
  - Study Site - 25008, Nantes, Loire Antlantique
  - Study Site - 25002, Paris, Paris
  - Study Site - 25004, Pau, Pyrenees Atlantiques
  - Study Site - 25001, Paris
- Germany (11):
  - Study Site 17001, Freiburg im Breisgau, Baden-Wurttemberg
  - Study Site 17005, Berlin, Berin
  - Study Site 17014, Franfurt, Hesse
  - Study Site 17012, Hanover, Lower Saxony
  - Study Site 17007, Lüdenscheid, North Rhine-Westphalia
  - Study Site 17010, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Study Site 17011, Mainz, Rhineland-Palatinate
  - Study Site 17003, Berlin
  - Study Site 17009, Berlin
  - Study Site 17002, Berlin
  - Study Site 17006, Hamburg
- Hungary (8):
  - Study Site 18008, Budapest
  - Study Site 18001, Budapest
  - Study Site 18005, Budapest
  - Study Site 18002, Győr
  - Study Site 18007, Nyíregyháza
  - Study Site 18003, Pécs
  - Study Site 18009, Szeged
  - Study Site 18006, Szolnok
- Israel (9):
  - Study Site 19010, Ashkelon
  - Study Site 19006, Beersheba
  - Study Site 19005, Haifa
  - Study Site 19004, Holon
  - Study Site 19003, Jerusalem
  - Study Site 19007, Jerusalem
  - Study Site 19002, Nahariya
  - Study Site 19009, Ramat Gan
  - Study Site 19008, Safed
- Italy (9):
  - Study Site 20003, Legnano, Milano
  - Study Site 20002, Magenta, Milano
  - Study Site 20008, Rozzano, Milano
  - Study Site 20009, Benevento
  - Study Site 20011, Napoli
  - Study Site 20007, Rimini
  - Study Site 20012, Roma
  - Study Site 20001, Terni
  - Study Site 20006, Udine
- Netherlands (12):
  - Study Site 21001, Alkmaar
  - Study Site 21006, Amsterdam
  - Study Site 21013, Amsterdam
  - Study Site 21016, Amsterdam
  - Study Site 21004, Ede
  - Study Site 21014, Leeuwarden
  - Study Site 21003, Nieuwegein
  - Study Site 21008, Nijmegen
  - Study Site 21009, Rotterdam
  - Study Site 21010, Sneek
  - Study Site 21015, Tilburg
  - Study Site 21011, Venlo
- Poland (11):
  - Study Site - 22015, Gdansk
  - Study Site - 22010, Grodzisk Mazowiecki
  - Study Site - 22012, Inowrocław
  - Study Site 22009, Kielce
  - Study Site - 22007, Krakow
  - Study Site - 22014, Lodz
  - Study Site - 22013, Starogard Gdański
  - Study Site - 22008, Warsaw
  - Study Site - 22006, Wałbrzych
  - Study Site - 22016, Wejherowo
  - Study Site - 22005, Wroclaw
- Spain (12):
  - Study Site - 23010, L'Hospitalet de Llobregat, Barcelona
  - Study Site - 23012, A Coruña, La Coruna
  - Study Site - 23006, Santiago de Compostela, La Coruna
  - Study Site - 23005, Barcelona
  - Study Site - 23002, Barcelona
  - Study Site - 23001, Barcelona
  - Study Site - 23003, Madrid
  - Study Site - 23013, Madrid
  - Study Site - 23004, Madrid
  - Study Site - 23007, Málaga
  - Study Site - 23009, Tarragona
  - Study Site - 23011, Valencia
- United Kingdom (6):
  - Study Site - 24006, Clydebank, Dunbartonshire
  - Study Site - 24004, Basildon, Essex
  - Study Site 24005, Romford, Essex
  - Study Site - 24003, London, Greater London
  - Study Site - 24010, Leicester, Leicestershire
  - Study Site - 24009, Newcastle upon Tyne, Tyne & Wear

REFERENCES:
- [Derived] Didichenko SA, Velkoska E, Navdaev AV, Greene BH, Lorkowski SW, Duffy D, Mears SJ, Wright SD, Gibson CM, Smith JD, Kingwell BA. CSL112 Infusion Rapidly Increases APOA1 Exchange Rate via Specific Serum Amyloid-Poor HDL Subpopulations When Administered to Patients Post-Myocardial Infarction. Arterioscler Thromb Vasc Biol. 2023 Jun;43(6):855-869. doi: 10.1161/ATVBAHA.122.318243. Epub 2023 Mar 30. PMID 36994730
- [Derived] Zheng B, Duffy D, Tricoci P, Kastrissios H, Pfister M, Wright SD, Gille A, Tortorici MA. Pharmacometric analyses to characterize the effect of CSL112 on apolipoprotein A-I and cholesterol efflux capacity in acute myocardial infarction patients. Br J Clin Pharmacol. 2021 Jun;87(6):2558-2571. doi: 10.1111/bcp.14666. Epub 2020 Dec 23. PMID 33217027
- [Derived] Michael Gibson C, Korjian S, Tricoci P, Daaboul Y, Yee M, Jain P, Alexander JH, Steg PG, Lincoff AM, Kastelein JJ, Mehran R, D'Andrea DM, Deckelbaum LI, Merkely B, Zarebinski M, Ophuis TO, Harrington RA. Safety and Tolerability of CSL112, a Reconstituted, Infusible, Plasma-Derived Apolipoprotein A-I, After Acute Myocardial Infarction: The AEGIS-I Trial (ApoA-I Event Reducing in Ischemic Syndromes I). Circulation. 2016 Dec 13;134(24):1918-1930. doi: 10.1161/CIRCULATIONAHA.116.025687. Epub 2016 Nov 15. PMID 27881559
- [Derived] Gibson CM, Korjian S, Tricoci P, Daaboul Y, Alexander JH, Steg PG, Lincoff AM, Kastelein JJ, Mehran R, D'Andrea D, Merkely B, Zarebinski M, Ophius TO, Harrington RA. Rationale and design of Apo-I Event Reduction in Ischemic Syndromes I (AEGIS-I): A phase 2b, randomized, placebo-controlled, dose-ranging trial to investigate the safety and tolerability of CSL112, a reconstituted, infusible, human apoA-I, after acute myocardial infarction. Am Heart J. 2016 Oct;180:22-8. doi: 10.1016/j.ahj.2016.06.017. Epub 2016 Jul 5. PMID 27659879

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Lead-in [CSL112 (2 g)]: In the safety lead-in, a small number of subjects (evenly stratified between subjects with normal renal function or mild renal impairment) were administered a single, 2 g infusion of CSL112.
- CSL112 (2 g): CSL112 (2 g) is to be administered as an intravenous (IV) infusion once weekly for 4 consecutive weeks.
  CSL112: CSL112 is a novel formulation of apolipoprotein A-I (apoA-I) purified from human plasma and reconstituted to form high-density lipoprotein (HDL) particles.
- CSL112 (6 g): CSL112 (6 g) is to be administered as an IV infusion once weekly for 4 consecutive weeks.
  CSL112: CSL112 is a novel formulation of apolipoprotein A-I (apoA-I) purified from human plasma and reconstituted to form high-density lipoprotein (HDL) particles.
Period: Overall Study
Arm/Group | Safety Lead-in [CSL112 (2 g)] | CSL112 (2 g) | CSL112 (6 g) | Placebo
Started | 9 | 419 | 421 | 418
Completed | 9 | 375 | 379 | 376
Not Completed | 0 | 44 | 42 | 42
Not completed — Non-compliance | 0 | 2 | 1 | 1
Not completed — Randomized by error/screen failure | 0 | 0 | 1 | 0
Not completed — Distance to center | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 11 | 6 | 12
Not completed — Death | 0 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 3 | 4
Not completed — Due to key hepatic values | 0 | 1 | 0 | 0
Not completed — Unable to contact patient | 0 | 3 | 1 | 2
Not completed — Patient unable to come to site/attend visit | 0 | 6 | 11 | 6
Not completed — Patient did not want another infusion | 0 | 3 | 3 | 2
Not completed — Vacation | 0 | 1 | 0 | 0
Not completed — Patient decision | 0 | 7 | 9 | 14
Not completed — Missed IV due to pharmacy error | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Lead-in [CSL112 (2 g)] | CSL112 (2 g) | CSL112 (6 g) | Placebo | Total
Number analyzed (Participants) | 9 | 419 | 421 | 418 | 1267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 306 | 296 | 301 | 910
  >=65 years | 2 | 113 | 125 | 117 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (7.19) | 57.7 (10.15) | 59.2 (9.87) | 58.1 (10.57) | 58.3 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 82 | 98 | 77 | 259
  Male | 7 | 337 | 323 | 341 | 1008
Region of Enrollment [Number; unit: participants]
  Hungary | 9 | 66 | 67 | 69 | 211
  United States | 0 | 59 | 54 | 54 | 167
  Czechia | 0 | 33 | 35 | 36 | 104
  United Kingdom | 0 | 3 | 2 | 4 | 9
  Spain | 0 | 6 | 5 | 6 | 17
  Canada | 0 | 9 | 9 | 7 | 25
  Austria | 0 | 2 | 3 | 2 | 7
  Netherlands | 0 | 48 | 48 | 49 | 145
  Denmark | 0 | 8 | 10 | 10 | 28
  Poland | 0 | 70 | 69 | 65 | 204
  Italy | 0 | 7 | 7 | 8 | 22
  Israel | 0 | 27 | 27 | 27 | 81
  Australia | 0 | 6 | 6 | 6 | 18
  Bulgaria | 0 | 47 | 47 | 46 | 140
  France | 0 | 0 | 2 | 1 | 3
  Germany | 0 | 28 | 30 | 28 | 86
Renal function from Interactive Web Response System (IWRS) [Number; unit: participants]
  Normal renal function | 4 | 195 | 192 | 191 | 582
  Mild renal impairment | 5 | 224 | 229 | 227 | 685

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Clinically Important Change in Drug-induced Liver Injury
Description: A clinically important change in drug-induced liver injury is defined as a change (from baseline) in alanine aminotransferase (ALT) greater than 3 times the upper limit of normal (ULN) or a change in total bilirubin greater than 2 times ULN, that is confirmed upon repeat measurement.
Time Frame: From baseline (before first infusion) to Day 29.
Population: The Safety population (SP) comprised all subjects who were randomized into the main study or PK/PD substudy and received at least a partial infusion of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 415 | 416 | 413
percentage of participants | 1.0 | 0.5 | 0
Statistical Analysis 1: Comparison: CSL112 (2 g) vs Placebo; Test type: Non-Inferiority — The calculation used a non-inferiority argument powering the test of the alternative hypothesis of no difference in the rates. Within each co-primary endpoint, the two active treatment groups are assumed to have the same endpoint rates. Total alpha is 0.05 with 0.025 allocated to each co-primary endpoint, which in turn involves comparisons of two active treatment groups to placebo without further alpha control; p = 0.1241, Newcombe-Wilson score method; Difference in event rates (%) = 1.0, 95% CI 2-sided [-0.1 to 2.5]
Statistical Analysis 2: Comparison: CSL112 (6 g) vs Placebo; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.4994, Newcombe-Wilson score method; Difference in event rates (%) = 0.5, 95% CI 2-sided [-0.5 to 1.7]

2. Primary Outcome: Percent of Participants With Clinically Important Change in Renal Status
Description: A clinically important change in renal status is defined as a serum creatinine (Cr) increase to ≥ 1.5 x the baseline value that is confirmed upon repeat measurement.
Time Frame: From baseline (before first infusion) to Day 29.
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 415 | 416 | 413
percentage of participants | 0 | 0.7 | 0.2
Statistical Analysis 1: Comparison: CSL112 (2 g) vs Placebo; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.4988, Newcombe-Wilson score method; Difference in event rates (%) = -0.2, 95% CI 2-sided [-1.4 to 0.7]
Statistical Analysis 2: Comparison: CSL112 (6 g) vs Placebo; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.6241, Newcombe-Wilson score method; Difference in event rates (%) = 0.5, 95% CI 2-sided [-0.7 to 1.9]

3. Secondary Outcome: The Percentage of Participants With a Time-to-first Major Adverse Cardiovascular Event (MACE)
Description: The MACE is a 4-component composite comprised of the time to the first of the following events: CV death, nonfatal myocardial infarction, ischemic stroke (non-hemorrhagic), and hospitalization for unstable angina.
Time Frame: From the start of the first infusion up to approximately 382 days
Population: The Intent-to-Treat (ITT) population comprised all subjects who were randomized to one of the three treatment groups for the Main Study or PK/PD substudy.
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 419 | 421 | 418
percentage of participants | 6.4 | 5.7 | 5.5
Statistical Analysis 1: Comparison: CSL112 (2 g) vs Placebo; Test type: Other; p = 0.5733, Log Rank — Stratified log-rank p-value; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.67 to 2.05]
Statistical Analysis 2: Comparison: CSL112 (6 g) vs Placebo; Test type: Other; p = 0.9717, Log Rank — Stratified log-rank p-value; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.57 to 1.80]

4. Secondary Outcome: Change From Baseline in Concentrations of Apolipoprotein A-I (apoA-I) and Phosphatidylcholine (PC) at End of First Infusion for All Participants
Description: Apolipoprotein A-I (apoA-I) and Phosphatidylcholine (PC) are analytes of CSL112
Time Frame: Before first infusion and end of first infusion
Population: The pharmacokinetic population (PK) comprised all subjects who received at least 1 infusion of investigational product and had at least 1 post baseline measurable plasma concentration of apoA-I or PC.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 396 | 404 | 403
mg/dL
  apoA-I | 35.9 (22.13) | 136.1 (54.37) | -4.7 (13.46)
  PC | 57.7 (31.12) | 180.4 (74.4) | -1.2 (20.43)

5. Secondary Outcome: Change From Baseline in Plasma Concentrations of apoA-I and PC at End of Fourth Infusion for All Participants
Time Frame: Before first infusion and end of fourth infusion
Population: PK
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 366 | 370 | 370
mg/dL
  apoA-I | 52.1 (55.03) | 158.0 (55.07) | 5.4 (26.47)
  PC | 48.7 (55.75) | 186.8 (79.39) | -12.9 (42.05)

6. Secondary Outcome: Change From Baseline in Plasma Concentrations of apoA-I and PC at End of First Infusion for Participants With Normal Renal Function
Description: apoA-I and PC are analytes of CSL112
Time Frame: Before first infusion and end of first infusion
Population: PK
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 185 | 175 | 183
mg/dL
  apoA-I | 36.0 (25.35) | 134.5 (48.25) | -4.0 (16.95)
  PC | 58.0 (37.06) | 177.4 (67.93) | -1.3 (25.74)

7. Secondary Outcome: Change From Baseline in Plasma Concentrations of apoA-I and PC at End of Fourth Infusion for Participants With Normal Renal Function
Description: apoA-I and PC are analytes of CSL112
Time Frame: Before first infusion and end of fourth infusion
Population: PK
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 173 | 160 | 171
mg/dL
  apoA-I | 54.7 (74.94) | 154.3 (53.64) | 4.8 (28.19)
  PC | 47.6 (64.67) | 182.0 (80.74) | -12.3 (44.89)

8. Secondary Outcome: Change From Baseline in Plasma Concentrations of apoA-I and PC at End of First Infusion for Participants With Mild Renal Impairment
Description: apoA-I and PC are analytes of CSL112
Time Frame: Before first infusion and end of first infusion
Population: PK
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 189 | 212 | 203
mg/dL
  apoA-I | 35.9 (19.05) | 135.5 (59.05) | -5.3 (9.7)
  PC | 57.8 (24.71) | 180.6 (79.50) | -0.8 (14.95)

9. Secondary Outcome: Change From Baseline in Plasma Concentrations of apoA-I and PC at End of Fourth Infusion for Participants With Mild Renal Impairment
Description: apoA-I and PC are analytes of CSL112
Time Frame: Before first infusion and end of fourth infusion
Population: PK
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 171 | 195 | 183
mg/dL
  apoA-I | 49.3 (27.63) | 158.4 (56.19) | 6.0 (25.68)
  PC | 50.6 (47.17) | 188.3 (79.39) | -13.2 (40.08)

10. Secondary Outcome: Change From Baseline in Plasma Cmax for apoA-I and PC After First Infusion for All Participants
Description: Cmax is the maximal plasma concentration.
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: The Pharmacokinetic/Pharmacodynamic (PK/PD) population was a subset of subjects from the main study who consented to participate in the PK/PD substudy.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 24 | 21 | 18
mg/dL
  apoA-I | 42.6 (11.2) | 147.4 (31.9) | 7.1 (7.9)
  PC | 67.7 (19.2) | 196.4 (36.2) | 11.1 (15.2)

11. Secondary Outcome: Change From Baseline in Plasma Cmax for apoA-I and PC After Fourth Infusion for All Participants
Description: Cmax is the maximal plasma concentration.
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 22 | 19 | 17
mg/dL
  apoA-I | 57.6 (19.5) | 164.3 (33.4) | 12.7 (19.5)
  PC | 59.0 (34.2) | 187.4 (49.9) | 9.1 (43.1)

12. Secondary Outcome: Change From Baseline in Plasma Cmax for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Description: Cmax is the maximal plasma concentration.
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 13 | 10 | 13
mg/dL
  apoA-I | 40.9 (12.0) | 135.1 (22.8) | 7.8 (8.3)
  PC | 61.9 (21.0) | 184.9 (31.5) | 13.0 (16.5)

13. Secondary Outcome: Change From Baseline in Plasma Cmax for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Description: Cmax is the maximal plasma concentration.
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 12 | 8 | 12
mg/dL
  apoA-I | 60.8 (19.2) | 149.0 (26.9) | 17.5 (20.3)
  PC | 45.8 (26.4) | 176.1 (54.0) | 20.1 (44.2)

14. Secondary Outcome: Change From Baseline in Plasma Cmax for apoA-I and PC After First Infusion for Participants With Mild Renal Impairment
Description: Cmax is the maximal plasma concentration.
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 11 | 10 | 5
mg/dL
  apoA-I | 44.6 (10.2) | 160.7 (37.0) | 5.2 (7.3)
  PC | 74.6 (14.7) | 211.3 (37.5) | 6.0 (10.8)

15. Secondary Outcome: Change From Baseline in Plasma Cmax for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Description: Cmax is the maximal plasma concentration.
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 10 | 5
mg/dL
  apoA-I | 53.7 (20.1) | 169.7 (29.3) | 1.0 (12.1)
  PC | 74.8 (37.0) | 190.4 (46.7) | -17.4 (28.9)

16. Secondary Outcome: Change From Baseline in Plasma Tmax for apoA-I and PC After First Infusion for All Participants
Description: Tmax is time to maximal plasma concentration
Time Frame: Before and for 7 days after the first infusion
Population: PK/PD
Measure: Median (Full Range); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 24 | 21 | 18
hours
  apoA-I | 2.23 [1.7 to 236.9] | 2.17 [2 to 4] | 46.8 [0 to 216.3]
  PC | 2.23 [1.7 to 8.4] | 2.17 [2 to 4] | 5.29 [0 to 188.9]

17. Secondary Outcome: Change From Baseline in Plasma Tmax for apoA-I and PC After Fourth Infusion for All Participants
Description: Tmax is time to maximal plasma concentration
Time Frame: Before and for 7 days after the fourth infusion
Population: PK/PD
Measure: Median (Full Range); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 22 | 19 | 17
hours
  apoA-I | 2.13 [2 to 23.5] | 2.25 [2 to 4.2] | 119 [0 to 332.9]
  PC | 2.17 [2 to 53.1] | 2.25 [2 to 4.2] | 46.93 [0 to 187.3]

18. Secondary Outcome: Change From Baseline in Plasma Tmax for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Description: Tmax is time to maximal plasma concentration
Time Frame: Before and for 7 days after the first infusion
Population: PK/PD
Measure: Median (Full Range); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 13 | 10 | 13
hours
  apoA-I | 2.25 [1.7 to 236.9] | 2.17 [2 to 3.4] | 96.1 [0 to 216.3]
  PC | 2.22 [1.7 to 8.4] | 2.17 [2 to 3.4] | 8.1 [0 to 188.9]

19. Secondary Outcome: Change From Baseline in Plasma Tmax for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Description: Tmax is time to maximal plasma concentration
Time Frame: Before and for 7 days after the fourth infusion
Population: PK/PD
Measure: Median (Full Range); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 12 | 8 | 12
hours
  apoA-I | 2.13 [2.1 to 3.5] | 2.17 [2 to 2.4] | 119.3 [0 to 332.9]
  PC | 2.17 [2.1 to 53.1] | 2.17 [2 to 2.4] | 29 [0 to 187.3]

20. Secondary Outcome: Change From Baseline in Plasma Tmax for apoA-I and PC After First Infusion for Participants With Mild Renal Impairment
Description: Tmax is time to maximal plasma concentration
Time Frame: Before and for 7 days after the first infusion
Population: PK/PD
Measure: Median (Full Range); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 11 | 10 | 5
hours
  apoA-I | 2.18 [2.1 to 3.4] | 2.22 [2.1 to 4] | 0 [0 to 117.9]
  PC | 2.28 [2.1 to 5] | 2.22 [2.1 to 4] | 0 [0 to 5.3]

21. Secondary Outcome: Change From Baseline in Plasma Tmax for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Description: Tmax is time to maximal plasma concentration
Time Frame: Before and for 7 days after the fourth infusion
Population: PK/PD
Measure: Median (Full Range); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 10 | 5
hours
  apoA-I | 2.17 [2 to 23.5] | 2.25 [2.1 to 4.2] | 72.5 [0 to 166.5]
  PC | 2.17 [2 to 8] | 2.25 [2.1 to 4.2] | 48.3 [9 to 166.5]

22. Secondary Outcome: Change From Baseline in Plasma Area Under the Curve (AUC) AUC0 - Last for apoA-I and PC After First Infusion for All Participants
Description: Area under the plasma concentration time curve (AUC) from time point zero (baseline) to the last quantifiable time-point before the analyte first returns to baseline [AUC0 - last]
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 24 | 21 | 18
mg•h/dL
  apoA-I | 1703 (2149) | 4819 (2580) | -766 (2248)
  PC | -66.12 (3653) | 869 (3796) | -2096 (3372)

23. Secondary Outcome: Change From Baseline in Plasma AUC0 - Last for apoA-I and PC After Fourth Infusion for All Participants
Description: as for outcome 22
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 22 | 19 | 17
mg•h/dL
  apoA-I | 4579 (2705) | 8985 (4263) | 747 (3226)
  PC | 70.7 (5327) | 2499 (7662) | -2185 (5189)

24. Secondary Outcome: Change From Baseline in Plasma AUC0 - Last for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Description: as for outcome 22
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 13 | 10 | 13
mg•h/dL
  apoA-I | 1278 (1742) | 3762 (2367) | -516 (2091)
  PC | -1382 (2853) | -137 (4057) | -1337 (2590)

25. Secondary Outcome: Change From Baseline in Plasma AUC0 - Last for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Description: as for outcome 22
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 12 | 8 | 12
mg•h/dL
  apoA-I | 4513 (2701) | 8609 (4500) | 1632 (3235)
  PC | -2130 (4691) | 3609 (10232) | -542 (4480)

26. Secondary Outcome: Change From Baseline in Plasma AUC0 - Last for apoA-I and PC After First Infusion for Subjects With Mild Renal Impairment
Description: as for outcome 22
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 11 | 10 | 5
mg•h/dL
  apoA-I | 2205 (2543) | 5917 (2568) | -1416 (2763)
  PC | 1489 (4003) | 1828 (3661) | -4068 (4634)

27. Secondary Outcome: Change From Baseline in Plasma AUC0 - Last for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Description: as for outcome 22
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 10 | 5
mg•h/dL
  apoA-I | 4659 (2854) | 8786 (4201) | -1376 (2205)
  PC | 2712 (5010) | 1541 (5815) | -6128 (4998)

28. Secondary Outcome: Change From Baseline in Plasma AUC0-t for apoA-I and PC After First Infusion for All Participants
Description: AUC from baseline to time point t (AUC0-t)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 24 | 21 | 18
mg•h/dL
  apoA-I (0-24h) | 496 (212) | 1929 (557) | -168 (158)
  apoA-I (0-48h) | 731 (447) | 2903 (944) | -331 (375)
  apoA-I (0-72h) | 880 (726) | 3516 (1248) | -439 (632)
  apoA-I (0-96h): number analyzed (Participants) | 24 | 20 | 18
  apoA-I (0-96h) | 1006 (1104) | 3943 (1581) | -541 (940)
  apoA-I (0-168h): number analyzed (Participants) | 16 | 20 | 10
  apoA-I (0-168h) | 1009 (1761) | 4734 (2382) | -452 (1498)
  PC (0-24h) | 508 (349) | 1545 (552) | -92 (229)
  PC (0-48h) | 466 (744) | 1627 (872) | -315 (522)
  PC (0-72h) | 418 (1251) | 1713 (1209) | -549 (886)
  PC (0-96h): number analyzed (Participants) | 23 | 21 | 18
  PC (0-96h) | 389 (1841) | 1712 (1694) | -780 (1346)
  PC (0-168h): number analyzed (Participants) | 16 | 15 | 11
  PC (0-168h) | -405 (3636) | 1273 (2764) | -1494 (2501)

29. Secondary Outcome: Change From Baseline in Plasma AUC0-t for apoA-I and PC After Fourth Infusion for All Participants
Description: AUC from baseline to time point t (AUC0-t)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 22 | 19 | 17
mg•h/dL
  apoA-I (0-24h) | 881 (422) | 2392 (655) | -57 (377)
  apoA-I (0-48h) | 1593 (798) | 3913 (1235) | -55 (759)
  apoA-I (0-72h) | 2195 (1177) | 5050 (1794) | -6 (1160)
  apoA-I (0-96h) | 2741 (1526) | 6000 (2292) | 90 (1590)
  apoA-I (0-168h): number analyzed (Participants) | 18 | 16 | 8
  apoA-I (0-168h) | 3997 (2655) | 8865 (3200) | 1635 (3540)
  PC (0-24h) | 462 (681) | 1564 (1051) | -488 (772)
  PC (0-48h) | 472 (1293) | 1765 (1948) | -902 (1433)
  PC (0-72h) | 509 (1989) | 1899 (2823) | -1173 (2168)
  PC (0-96h) | 518 (2679) | 1951 (3681) | -1417 (2894)
  PC (0-168h): number analyzed (Participants) | 16 | 16 | 8
  PC (0-168h) | -625 (4963) | 2655 (6024) | -442 (6319)

30. Secondary Outcome: Change From Baseline in Plasma AUC0-t for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Description: AUC from baseline to time point t (AUC0-t)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 13 | 10 | 13
mg•h/dL
  apoA-I (0-24h) | 418 (117) | 1653 (496) | -149 (123)
  apoA-I (0-48h) | 547 (204) | 2521 (955) | -316 (332)
  apoA-I (0-72h) | 628 (337) | 3064 (1280) | -435 (579)
  apoA-I (0-96h): number analyzed (Participants) | 13 | 9 | 13
  apoA-I (0-96h) | 692 (554) | 3342 (1642) | -528 (883)
  apoA-I (0-168h): number analyzed (Participants) | 8 | 9 | 7
  apoA-I (0-168h) | 821 (1387) | 3780 (2353) | -275 (1461)
  PC (0-24h) | 364 (245) | 1347 (661) | -46 (160)
  PC (0-48h) | 145 (536) | 1294 (1025) | -235 (441)
  PC (0-72h) | -38 (946) | 1325 (1421) | -426 (759)
  PC (0-96h) | -256 (1415) | 1218 (2005) | -569 (1162)
  PC (0-168h): number analyzed (Participants) | 9 | 7 | 7
  PC (0-168h) | -1511 (3053) | 437 (2061) | -1089 (2188)

31. Secondary Outcome: Change From Baseline in Plasma AUC0-t for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Description: AUC from baseline to time point t (AUC0-t)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 12 | 8 | 12
mg•h/dL
  apoA-I (0-24h) | 929 (396) | 2098 (463) | 20 (417)
  apoA-I (0-48h) | 1668 (753) | 3459 (1001) | 105 (820)
  apoA-I (0-72h) | 2252 (1116) | 4497 (1478) | 249 (1232)
  apoA-I (0-96h) | 2769 (1473) | 5360 (1909) | 459 (1666)
  apoA-I (0-168h): number analyzed (Participants) | 10 | 6 | 7
  apoA-I (0-168h) | 3811 (2706) | 8342 (2549) | 2486 (2804)
  PC (0-24h) | 189 (483) | 1524 (1388) | -295 (819)
  PC (0-48h) | -59 (952) | 1796 (2613) | -523 (1446)
  PC (0-72h) | -306 (1544) | 2000 (3773) | -605 (2133)
  PC (0-96h) | -573 (2204) | 2078 (4905) | -633 (2772)
  PC (0-168h): number analyzed (Participants) | 8 | 6 | 7
  PC (0-168h) | -3853 (3242) | 4584 (7822) | 1253 (4446)

32. Secondary Outcome: Change From Baseline in Plasma AUC0-t for apoA-I and PC After First Infusion for Participants With Mild Renal Impairment
Description: AUC from baseline to time point t (AUC0-t)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 11 | 10 | 5
mg•h/dL
  apoA-I (0-24h) | 589 (263) | 2219 (515) | -218 (238)
  apoA-I (0-48h) | 949 (560) | 3308 (847) | -370 (514)
  apoA-I (0-72h) | 1179 (946) | 3998 (1152) | -451 (834)
  apoA-I (0-96h) | 1376 (1468) | 4517 (1465) | -576 (1188)
  apoA-I (0-168h): number analyzed (Participants) | 8 | 10 | 3
  apoA-I (0-168h) | 1196 (2155) | 5624 (2293) | -865 (1824)
  PC (0-24h) | 678 (386) | 1777 (353) | -212 (348)
  PC (0-48h) | 845 (797) | 1968 (623) | -523 (705)
  PC (0-72h) | 956 (1393) | 2093 (950) | -871 (1196)
  PC (0-96h): number analyzed (Participants) | 10 | 10 | 5
  PC (0-96h) | 1227 (2058) | 2194 (1351) | -1329 (1769)
  PC (0-168h): number analyzed (Participants) | 7 | 8 | 4
  PC (0-168h) | 1018 (4052) | 2004 (3214) | 2203 (3197)

33. Secondary Outcome: Change From Baseline in Plasma AUC0-t for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Description: AUC from baseline to time point t (AUC0-t)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 10 | 5
mg•h/dL
  apoA-I (0-24h) | 823 (466) | 2469 (573) | -243 (170)
  apoA-I (0-48h) | 1503 (881) | 4049 (1221) | -440 (436)
  apoA-I (0-72h) | 2128 (1304) | 5226 (1910) | -617 (741)
  apoA-I (0-96h) | 2707 (1669) | 6212 (2503) | -796 (1045)
  apoA-I (0-168h): number analyzed (Participants) | 8 | 9 | 1
  apoA-I (0-168h) | 4229 (2754) | 8840 (3678) | -4322 (0)
  PC (0-24h) | 789 (760) | 1518 (799) | -950 (405)
  PC (0-48h) | 1110 (1402) | 1650 (1474) | -1810 (1001)
  PC (0-72h) | 1487 (2090) | 1726 (2176) | -2536 (1731)
  PC (0-96h) | 1826 (2706) | 1751 (2867) | -3297 (2471)
  PC (0-168h): number analyzed (Participants) | 8 | 9 | 1
  PC (0-168h) | 2603 (4295) | 1316 (4998) | -12308 (0)

34. Secondary Outcome: Change From Baseline in Plasma AUC0-∞ for apoA-I and PC After First Infusion for All Participants
Description: AUC0-∞ is plasma area under the curve (AUC0-infinity)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 6 | 16 | 1
mg•h/dL
  apoA-I: number analyzed (Participants) | 6 | 16 | 0
  apoA-I | 1425 (1297) | 6090 (3642) |
  PC: number analyzed (Participants) | 6 | 10 | 1
  PC | 1850 (3120) | 1678 (651) | 6979 (0)

35. Secondary Outcome: Change From Baseline in Plasma AUC0-∞ for apoA-I and PC After Fourth Infusion for All Participants
Description: AUC0-∞ is plasma area under the curve (AUC0-infinity)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 15 | 1
mg•h/dL
  apoA-I | 15540 (19437) | 13570 (6965) | 4615 (0)
  PC: number analyzed (Participants) | 6 | 11 | 0
  PC | 2015 (2855) | 12863 (16731) |

36. Secondary Outcome: Change From Baseline in Plasma AUC0-∞ for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Description: AUC0-∞ is plasma area under the curve (AUC0-infinity)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 3 | 8 | 0
mg•h/dL
  apoA-I: number analyzed (Participants) | 2 | 8 | 0
  apoA-I | 589 (17) | 4505 (2528) |
  PC: number analyzed (Participants) | 3 | 5 | 0
  PC | 490 (1540) | 1596 (785) |

37. Secondary Outcome: Change From Baseline in Plasma AUC0-∞ for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Description: AUC0-∞ is plasma area under the curve (AUC0-infinity)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 7 | 5 | 1
mg•h/dL
  apoA-I | 17079 (23224) | 12422 (7399) | 4615 (0)
  PC: number analyzed (Participants) | 4 | 3 | 0
  PC | 638 (566) | 16142 (17777) |

38. Secondary Outcome: Change From Baseline in Plasma AUC0-∞ for apoA-I and PC After First Infusion for Participants With Mild Renal Impairment
Description: AUC0-∞ is plasma area under the curve (AUC0-infinity)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 4 | 7 | 1
mg•h/dL
  apoA-I: number analyzed (Participants) | 4 | 7 | 0
  apoA-I | 1842 (1451) | 8032 (4220) |
  PC: number analyzed (Participants) | 3 | 5 | 1
  PC | 3210 (4052) | 1761 (566) | 6979 (0)

39. Secondary Outcome: Change From Baseline in Plasma AUC0-∞ for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Description: AUC0-∞ is plasma area under the curve (AUC0-infinity)
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: mg•h/dL
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 3 | 9 | 0
mg•h/dL
  apoA-I | 11951 (7374) | 13157 (6734) |
  PC: number analyzed (Participants) | 2 | 7 | 0
  PC | 4769 (4128) | 12827 (18453) |

40. Secondary Outcome: Change From Baseline in Plasma Terminal Half-life (t1/2) for apoA-I and PC After First Infusion for All Participants
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 6 | 16 | 1
hours
  apoA-I: number analyzed (Participants) | 6 | 16 | 0
  apoA-I | 46.4 (33.1) | 53.9 (38.7) |
  PC: number analyzed (Participants) | 6 | 10 | 1
  PC | 32.9 (29.6) | 9.7 (7.2) | 241.2 (0)

41. Secondary Outcome: Change From Baseline in Plasma Terminal Half-life (t1/2) for apoA-I and PC After Fourth Infusion for All Participants
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 15 | 1
hours
  apoA-I | 269.1 (292) | 103.6 (61.1) | 145 (0)
  PC: number analyzed (Participants) | 6 | 11 | 0
  PC | 21.5 (20.6) | 156.3 (245.8) |

42. Secondary Outcome: Change From Baseline in Plasma Terminal Half-life (t1/2) for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 3 | 8 | 0
hours
  apoA-I: number analyzed (Participants) | 2 | 8 | 0
  apoA-I | 7.5 (1.7) | 41.4 (24.1) |
  PC: number analyzed (Participants) | 3 | 5 | 0
  PC | 34 (27.7) | 12.3 (8.9) |

43. Secondary Outcome: Change From Baseline in Plasma Terminal Half-life (t1/2) for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 7 | 5 | 1
hours
  apoA-I | 271.6 (317.4) | 96.5 (47.3) | 145 (0)
  PC: number analyzed (Participants) | 4 | 3 | 0
  PC | 9.1 (9.3) | 121.1 (102.7) |

44. Secondary Outcome: Change From Baseline in Plasma Terminal Half-life (t1/2) for apoA-I and PC After First Infusion for Participants With Mild Renal Impairment
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 4 | 7 | 1
hours
  apoA-I: number analyzed (Participants) | 4 | 7 | 0
  apoA-I | 65.9 (17.5) | 66.4 (51.4) |
  PC: number analyzed (Participants) | 3 | 5 | 1
  PC | 31.8 (37.7) | 7.1 (4.4) | 241.2 (0)

45. Secondary Outcome: Change From Baseline in Plasma Terminal Half-life (t1/2) for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 3 | 9 | 0
hours
  apoA-I | 263.1 (285.4) | 99.2 (68.2) |
  PC: number analyzed (Participants) | 2 | 7 | 0
  PC | 46.3 (2.2) | 185.6 (306.5) |

46. Secondary Outcome: Change From Baseline in Plasma Clearance (CL) for apoA-I and PC After First Infusion for All Participants
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 6 | 16 | 0
L/h
  apoA-I | 0.29 (0.27) | 0.15 (0.13) |
  PC: number analyzed (Participants) | 5 | 10 | 0
  PC | 0.32 (0.26) | 0.61 (0.26) |

47. Secondary Outcome: Change From Baseline in Plasma Clearance (CL) for apoA-I and PC After Fourth Infusion for All Participants
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 17 | 16 | 0
L/h
  apoA-I | 0.09 (0.1) | 0.07 (0.02) |
  PC: number analyzed (Participants) | 6 | 11 | 0
  PC | 0.11 (0.09) | 0.57 (1.12) |

48. Secondary Outcome: Change From Baseline in Plasma Clearance (CL) for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 2 | 8 | 0
L/h
  apoA-I | 0.33 (0.01) | 0.19 (0.17) |
  PC: number analyzed (Participants) | 2 | 5 | 0
  PC | 0.41 (0.38) | 0.68 (0.35) |

49. Secondary Outcome: Change From Baseline in Plasma Clearance (CL) for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 6 | 0
L/h
  apoA-I | 0.11 (0.12) | 0.08 (0.02) |
  PC: number analyzed (Participants) | 1 | 5 | 0
  PC | 0.24 (0) | 0.19 (0.12) |

50. Secondary Outcome: Change From Baseline in Plasma Clearance (CL) for apoA-I and PC After First Infusion for Participants With Mild Renal Impairment
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 4 | 7 | 0
L/h
  apoA-I | 0.27 (0.35) | 0.09 (0.05) |
  PC: number analyzed (Participants) | 3 | 5 | 0
  PC | 0.26 (0.23) | 0.54 (0.13) |

51. Secondary Outcome: Change From Baseline in Plasma Clearance (CL) for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 7 | 9 | 0
L/h
  apoA-I | 0.05 (0.02) | 0.08 (0.03) |
  PC: number analyzed (Participants) | 5 | 5 | 0
  PC | 0.08 (0.07) | 1.01 (1.63) |

52. Secondary Outcome: Change From Baseline in Plasma Volume of Distribution at Steady State (Vss) for apoA-I and PC After First Infusion for All Participants
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 6 | 16 | 0
Liters
  apoA-I | 33.4 (64.7) | 7.4 (3.1) |
  PC: number analyzed (Participants) | 5 | 10 | 0
  PC | 6.1 (4.4) | 14.4 (33.3) |

53. Secondary Outcome: Change From Baseline in Plasma Vss for apoA-I and PC After Fourth Infusion for All Participants
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 10 | 15 | 0
Liters
  apoA-I | 18.7 (16.6) | 9.4 (4.7) |
  PC: number analyzed (Participants) | 6 | 11 | 0
  PC | 10.7 (7.5) | 58.3 (94.9) |

54. Secondary Outcome: Change From Baseline in Plasma Vss for apoA-I and PC After First Infusion for Participants With Normal Renal Function
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 2 | 8 | 0
Liters
  apoA-I | 3.8 (0.9) | 8.1 (3.8) |
  PC: number analyzed (Participants) | 2 | 5 | 0
  PC | 8.3 (7.7) | 24.7 (47.2) |

55. Secondary Outcome: Change From Baseline in Plasma Vss for apoA-I and PC After Fourth Infusion for Participants With Normal Renal Function
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 7 | 5 | 0
Liters
  apoA-I | 18.7 (16.1) | 9.4 (2.5) |
  PC: number analyzed (Participants) | 4 | 3 | 0
  PC | 11.4 (8.3) | 17 (10.3) |

56. Secondary Outcome: Change From Baseline in Plasma Vss for apoA-I and PC After First Infusion for Participants With Mild Renal Impairment
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after first infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 4 | 7 | 0
Liters
  apoA-I | 48.2 (78.1) | 6.4 (2.3) |
  PC: number analyzed (Participants) | 3 | 5 | 0
  PC | 4.7 (1.3) | 4 (1.5) |

57. Secondary Outcome: Change From Baseline in Plasma Vss for apoA-I and PC After Fourth Infusion for Participants With Mild Renal Impairment
Time Frame: Before first infusion (baseline) and for up to approximately 7 days after fourth infusion
Population: PK/PD
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 3 | 9 | 0
Liters
  apoA-I | 18.7 (21.3) | 9.4 (5.9) |
  PC: number analyzed (Participants) | 2 | 7 | 0
  PC | 9.3 (8.2) | 83.1 (114) |

58. Secondary Outcome: Percent of Participants With the Occurrence of Suspected Adverse Drug Reactions
Description: The overall percentage of subjects:
  * with adverse events (AEs), including local tolerability events, that begin during or within 1 hour of an infusion; or
  * with AEs considered to be causally related to the test product; or
  * who experience an AE for which the incidence rate in an active treatment arm exceeds the exposure-adjusted incidence rate in the placebo arm by 30% or more, provided the difference in incidence rates is 1% or more.
Time Frame: From the start of first infusion, up to approximately Day 382
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 415 | 416 | 413
percentage of participants | 31.8 | 28.4 | 23.5

59. Secondary Outcome: Percent of Participants With Any Adverse Event (AE)
Time Frame: From the start of first infusion, up to approximately Day 382
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 415 | 416 | 413
percentage of participants | 50.6 | 51.4 | 49.6

60. Secondary Outcome: Percent of Participants Who Experience Bleeding Events
Description: The number of subjects who experience bleeding events as defined by the Bleeding Academic Research Consortium (BARC) criteria (Mehran et al, 2011)
Time Frame: From the start of first infusion, up to approximately Day 112
Population: SP
Measure: Number; unit: percentage of participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 415 | 416 | 413
percentage of participants | 9.2 | 9.1 | 12.3

61. Secondary Outcome: Change From Baseline in Serum Antibodies to CSL112 and apoA-I
Time Frame: Before first infusion, up to approximately Day 112
Population: SP
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 377 | 389 | 380
Titer
  Anti-CSL112 antibody | 0 (0.14) | 0 (0.2) | 0 (0.2)
  Anti-apoA-I antibody | 0 (0.09) | 0 (0.14) | 0 (0.1)

62. Secondary Outcome: Number of Participants With Positive Serology Results for IgG and IgM Antibodies to Parvovirus B19
Time Frame: Study Day 112
Population: Serology population are a random subset of participants that was selected and had their samples tested for the presence of parvovirus B19.
Measure: Number; unit: participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 60 | 60 | 60
participants
  IgG | 40 | 48 | 44
  IgM | 0 | 0 | 0

63. Secondary Outcome: Number of Participants With Parvovirus B19 DNA in Serum
Time Frame: Study Day 112
Population: Serology population
Measure: Number; unit: participants
Arm/Group | CSL112 (2 g) | CSL112 (6 g) | Placebo
Number analyzed (Participants) | 60 | 60 | 60
participants
  Not detected | 57 | 60 | 59
  < 101 IU/mL | 1 | 0 | 1
  Missing | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 382 days for each participant
Groups:
- CSL112 (2 g): CSL112 (2 g) is to be administered as an intravenous (IV) infusion once weekly for 4 consecutive weeks.
- CSL112 (6 g): CSL112 (6 g) is to be administered as an IV infusion once weekly for 4 consecutive weeks.
Arm/Group | Safety Lead-in [CSL112 (2 g)] | CSL112 (2 g) | CSL112 (6 g) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/9 | 5/415 | 4/416 | 1/413
Serious Adverse Events (participants affected / at risk) | 1/9 | 66/415 | 54/416 | 55/413
Other Adverse Events (participants affected / at risk) | 2/9 | 15/415 | 23/416 | 9/413
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead-in [CSL112 (2 g)] (N=9) | CSL112 (2 g) (N=415) | CSL112 (6 g) (N=416) | Placebo (N=413)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 9 (10) | 4 (4) | 5 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 4 (4) | 4 (6)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular stent restenosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Vascular stent thrombosis (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 5 (5) | 6 (7) | 5 (6)
Angina unstable (Cardiac disorders) | 0 (0) | 6 (6) | 3 (3) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac asthma (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular septal defect acquired (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead-in [CSL112 (2 g)] (N=9) | CSL112 (2 g) (N=415) | CSL112 (6 g) (N=416) | Placebo (N=413)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 15 (19) | 23 (24) | 9 (10)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes